CLINICAL TRIAL: NCT06729138
Title: Resisted Training in Runners. A Randomized Controlled Trial.
Brief Title: Resisted Training in Runners
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cadiz (Other)
Responsible Party: Principal Investigator, Pablo Góngora Rodríguez, MSc in Research on Physical Activity and Sport, University of Cadiz
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: PGR0001
Record Dates: First submitted 2024-11-24; First posted 2024-12-11 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2024-10

CONDITIONS: Performance Enhancing
Keywords: Runners; Sprint; Performance; Sled training; Track and field
MeSH Terms: interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sprint training (Active Comparator)
  Interventions: Other: Sprint Training
- Resisted Sprint (Experimental)
  Interventions: Other: Resisted Sprint Training

INTERVENTIONS:
Other: Resisted Sprint Training — In this intervention, participants will perform 16 sessions of resisted sprint training with external loads using a sled over eight weeks. In these 16 sessions the intensity will vary in both the distance to be covered and the load to be moved.
  Arms: Resisted Sprint
Other: Sprint Training — In this intervention, participants will perform 16 sessions of sprint training over eight weeks. In these 16 sessions the intensity will vary in the distance.
  Arms: Sprint training

SUMMARY:
INTRODUCTION: Sprint training and resisted sprint training with sled has generated interest in the scientific literature due to its potential to improve performance, different studies have shown that incorporating strength training and sprints into studies have shown that the incorporation of strength and sprint training into the training programmes of long-distance runners can have significant training programmes for long-distance runners can have significant effects on running economy, anaerobic capacity of the runners and the anaerobic capacity of athletes, along with various neuromuscular adaptations. Despite these findings, the application of sprint and resisted sprint training with dragging in middle-distance and long-distance runners has been and long-distance runners has been scarcely studied, with most studies focusing on sprinters and athletes from team sports and sprinters, leaving a gap in the understanding of how these methods can influence distance runners. Along with how the intensity of external external loads affect this type of work and the influence on key kinetic variables such as vertical oscillation, contact time with the oscillation, ground contact time and muscle stiffness in this specific population.

PURPOSE: Analyse the effects that sprint training and resisted sprint training can have on running economy, force production, speed and various kinetics variables such as vertical oscillation, contact time, speed and vertical oscillation, ground contact time and muscle stiffness. MATERIAL AND METHODS: A randomised, longitudinal, prospective, blinded, assessor-blinded clinical trial will be conducted. Different variables related to sports performance will be evaluated, such as maximum oxygen consumption, critical power, heart rate variability or kinetic variables, among others.

kinetic variables among others. The evaluation will be carried out before the application of the training intervention and after two months. The study will be conducted with runners recruited through athletics clubs in the region of Cadiz, being randomly assigned a system of numerical tables using a computer programme between the sprint group (n=40) and the resisted sprint group (n=40). Both groups will perform two training sessions training sessions for eight weeks, consisting of sprint or resisted sprint repetitions based on the assigned group.

KEY WORDS: athletics, runners, resisted training, sprint.

ELIGIBILITY:
Inclusion Criteria:

* At least 2 years of training experience as a runner.
* Do more than 30 kilometres per week.
* Perform at least 3 training sessions per week.
* Have competed in a 10km race or longer distance in the last 6 months.
* Be between 18 and 35 years old.
* Availability to attend the proposed training sessions.

Exclusion Criteria:

* Have a musculoskeletal injury or have had a musculoskeletal injury in the 6 months prior to the start of the study.
* Have chronic diseases.
* Have a BMI over 24.9.
* Combine training and competition in other disciplines other than running.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-04-10 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
V02 max | Through study completion, an average of 10 weeks
  VO2 Max (Maximum Oxygen Consumption) is the maximum amount of oxygen that an individual can utilize during intense or maximal exercise. It is a key indicator of cardiovascular and aerobic fitness, reflecting the capacity of the heart, lungs, and muscles to deliver and use oxygen efficiently. VO2 Max is typically measured in milliliters of oxygen consumed per kilogram of body weight per minute (ml/kg/min). A higher VO2 Max value generally indicates better endurance performance.
Critical Power | Through study completion, an average of 10 weeks
  Critical power (CP) is the maximum work intensity that an athlete can maintain consistently over a prolonged period of time.
Jump Height | Through study completion, an average of 10 weeks. In each training sesion.
  This is the height reached in centimetres during the performance of the countermovement jump and the box jump.
  countermovement jump and jump from the box. Both tests and their respective jumping heights provide valuable information on the explosive and reactive strength capacity of the leg muscles.
Heart Rate | Through study completion, an average of 10 weeks
  Heart rate is measured in beats per minute (bpm) and is an important indicator of cardiovascular function and exercise intensity. The maximum heart rate is the maximum number of heartbeats the heart can achieve per minute during maximum physical exertion. It is an individual value, although there are different formulas for its calculation, it can vary significantly between trained and untrained individuals or by trained or untrained individuals or for other reasons.
Heart Rate Variability | Through study completion, an average of 10 weeks
  Heart Rate Variability (HRV) is the variation in the time intervals between consecutive heartbeats, measured in milliseconds. It reflects the ability of the autonomic nervous system (ANS) to adapt to changing physiological demands by balancing sympathetic ("fight or flight") and parasympathetic ("rest and digest") activity. A higher HRV typically indicates greater cardiovascular and nervous system adaptability, resilience, and recovery, while a lower HRV may signal stress, fatigue, or decreased fitness. HRV is often used as a marker for overall health, recovery, and readiness in both clinical and athletic contexts.
Stride Length | Through study completion, an average of 10 weeks
  Stride length is the distance a runner covers with each step during a run. It is measured from the point of contact of one foot to the point of contact of the same foot in the next step. It is a key metric in the biomechanics of running and can significantly influence a runner's performance and efficiency.
Vertical oscillation | Through study completion, an average of 10 weeks
  Vertical oscillation in the context of running biomechanics refers to the upward and downward movement of the body's centre of mass during the running cycle. This vertical motion is a natural component of the running movement pattern and It occurs as a result of the complex interaction between momentum forces and gait dynamics.
Contact time | Through study completion, an average of 10 weeks
  Contact time in biomechanical running terms refers to the period of time a runner's foot is in contact with the ground during each stride cycle.
Perceived exertion | In each training session through study completion, an average of 10 weeks
  Perceived exertion refers to an individual's subjective perception of the intensity or difficulty of a physical activity.
Body Mass Index (BMI) | Through study completion, an average of 10 weeks
  Body Mass Index (BMI) is a numerical value calculated by dividing a person's weight in kilograms by the square of their height in meters (kg/m²). It is a widely used screening tool to categorize individuals into weight categories such as underweight, normal weight, overweight, or obese, based on their body composition. Although BMI does not directly measure body fat percentage, it provides a general indication of whether a person's weight is appropriate for their height and is commonly used in public health and clinical settings.

CONTACTS AND LOCATIONS:
Locations (1):
- CD Atletismo Bahía de Cádiz, Cadiz, Andalusia, Spain

IPD SHARING:
Plan to Share IPD: Yes
All data about the study will be shared, while maintaining the confidentiality of the participants.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: All data will be available from the end of the study. And thereafter for a period of 10 years.
Access Criteria: Access to the data will be granted to all researchers who request it by the appropriate means and always respecting the confidentiality of the participants' data.